CLINICAL TRIAL: NCT06085521
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficiency and Safety of LNK01001 Capsule in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of LNK01001 Capsule in Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LK001202
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LNK01001 Dose A (Experimental): Participants will receive LNK01001capsule Dose A BID orally for 12 weeks.
  Interventions: Drug: LNK01001 Dose A
- LNK01001 Dose B (Experimental): Participants will receive LNK01001capsule Dose B BID orally for 12 weeks.
  Interventions: Drug: LNK01001 Dose B
- placebo (Placebo Comparator): Participants will receive a Placebo capsule BID orally for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LNK01001 Dose A — Capsules taken orally
  Arms: LNK01001 Dose A
Drug: LNK01001 Dose B — Capsules taken orally
  Arms: LNK01001 Dose B
Drug: placebo — Capsules taken orally
  Arms: placebo

SUMMARY:
Participants who meet eligibility criteria will be randomized in a 1:1:1 ratio to receive a twice daily oral LNK01001 dose A or LNK01001 dose B or matching placebo for 12 weeks.

DETAILED DESCRIPTION:
The study was to include a 12-week double-blind treatment period. Participants who met eligibility criteria were to be randomized in a 1:1:1 ratio to one of the three treatment groups.

Group 1:LNK01001 dose A (Day 1 to Week 12) Group 2:LNK01001 dose B (Day 1 to Week 12) Group 3: Matching placebo (Day 1 to Week 12)

ELIGIBILITY:
Inclusion Criteria:

* participants between ≥ 18 and ≤75 years of age.
* subjects meet Hanifin and Rajka criteria.
* subjects meet moderate to severe AD criteria.
* inadequate response to topical treatment or systemic treatment for AD within 6 months before screening.

Exclusion Criteria:

* current use of topical treatment for AD within 2 weeks before baseline visit.
* prior exposure to Janus Kinase (JAK) inhibitor.
* prior exposure to phototherapy, tanning bed, or any other light emitting device treatment within 4 weeks before baseline visit.
* Prior exposure to any Biologic treatment including Dupilumab, Omalizumab within 3 months before baseline visit.
* Any significant clinical and laboratory abnormalities, as determined by the Investigator, may affect the safety of the subjects, including but not limited to:WBC<3×10e9/L, neutrophil<1.2×10e9/L, platelet<100×10e9/L, hemoglobin<85 g/L; Aspartate aminotransferase or alanine aminotransferase>1.5×ULN, or total bilirubin>1.5×ULN; Serum creatinine>1.2×ULN.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Eczema Area and Severity Index (EASI) Score | week 12
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved a 75% Reduction in EASI Score (EASI 75) | Week 4,8,12
  An EASI 75 response is defined as participants with at least a 75% reduction (improvement) in EASI score relative to the Baseline value
Percentage of Participants Achieving an Investigator Global Assessment (IGA) response | Week 4,8,12
  IGA response defined as an IGA score of 0 (clear) or 1 (almost clear) with a reduction from baseline of ≥ 2 points
Percent Change from Baseline in EASI Score | Week 4,8
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percentage of Participants Achieving a Reduction of ≥ 3 Points From Baseline in Worst Pruritus Numerical Rating Scale (NRS) | Week 4,8,12
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Change From Baseline in Worst Pruritus Numerical Rating Scale(NRS) Score | Week 4,8,12
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Percentage of Participants Achieving a Reduction of ≥ 2 Points From Baseline in Investigator Global Assessment (IGA) | Week 4,8,12
  IGA is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  0 - Clear: No inflammatory signs of AD;
  1. - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  2. - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  3. - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  4. - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Percentage of Participants Who Achieved a 90% Reduction in EASI Score (EASI 90) | Week 4,8,12
  An EASI 90 response is defined as participants with at least a 90% reduction (improvement) in EASI score relative to the Baseline value
Percentage of Participants Who Achieved a 50% Reduction in EASI Score (EASI 50) | Week 4,8,12
  An EASI 50 response is defined as participants with at least a 50% reduction (improvement) in EASI score relative to the Baseline value
Percent Change from Baseline in Scoring Atopic Dermatitis (SCORAD) Score | Week 4,8,12
  SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst). A negative change from Baseline indicates improvement.
Change From Baseline in Dermatology Life Quality Index (DLQI) Score | Week 4,8,12
  The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL.
Change From Baseline in Patient Oriented Eczema Measure (POEM) Score | Week 4,8,12
  The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults. Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema). A change in POEM score of 3.4 points is considered the minimal clinically important difference.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Jianzhong Zhang, Beijing, China